CLINICAL TRIAL: NCT06982014
Title: The Effect of Simulation Training Using the Moulage Technique on Nursing Students' Knowledge and Attitudes Toward Identifying Physical Violence
Brief Title: Impact of Moulage-Based Simulation on Nursing Students' Recognition of Physical Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 150325
Record Dates: First submitted 2025-04-28; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Nursing Education
Keywords: Moulage-based simulation; Violence against women; Nursing education; Physical violence recognition; Educational methods
MeSH Terms: interventions — Models, Anatomic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The intervention applied to the experimental group involves moulage-based simulation training designed to enhance the recognition of physical violence against women. The process includes the following steps:
  Simulation Scenarios: Students in the experimental group will work with clinical simulation scenarios featuring cases with physical violence signs. These scenarios are specifically designed to improve students' ability to recognize the indicators of violence against women.
  Standardized Patient Modality: The experimental group will engage in simulated interactions with a standardized patient (moulage) who displays signs of violence. This allows students to realistically assess the physical signs of violence and practice their recognition skills.
  Training Process: Prior to the simulation, students will receive a briefing on how to recognize violence signs, including physical, sexual, emotional violence, and related health care services. This information will prepare them to effec
  Interventions: Behavioral: cilinical simulation
- control group (Active Comparator): The intervention process for the control group involves a more traditional educational approach, specifically focusing on raising awareness about gender-based violence through media and instructional materials. The process for the control group is as follows:
  Educational Video Viewing: The control group will watch a film titled "Gözlerimde Al" (translated as "Take My Eyes"), which addresses the issue of gender-based violence. The film aims to provide insights into the emotional and physical effects of violence against women and encourages reflection on how to recognize such violence in real-life scenarios.
  Pre-Training Assessment: Before the video viewing, the control group will complete a pre-training assessment, which includes a demographic data form and the ISKEBE Attitude Scale towards Violence Against Women. This assessment helps establish baseline knowledge and attitudes regarding gender-based violence.
  Post-Training Reflection: After watching the film, students in the contro
  Interventions: Other: Educational Video Viewing

INTERVENTIONS:
Behavioral: cilinical simulation — he experimental group will interact with standardized patients (using moulage techniques) who exhibit signs of physical violence. This approach provides a realistic environment for students to assess the physical manifestations of violence and practice their recognition skills in a controlled, yet lifelike, setting.
  Other Names: moulage
  Arms: experimental group
Other: Educational Video Viewing — The control group will watch a film titled "Gözlerimde Al" (translated as "Take My Eyes"), which addresses the issue of gender-based violence. The film aims to provide insights into the emotional and physical effects of violence against women and encourages reflection on how to recognize such violence in real-life scenarios.
  Arms: control group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of moulage-based simulation training in improving nursing students' ability to recognize physical violence in women. The main questions it aims to answer are:

Does moulage-based simulation improve nursing students' ability to recognize signs of physical violence in women compared to traditional training methods? How does the simulation affect nursing students' attitudes and knowledge about gender-based violence? Researchers will compare an experimental group, which will participate in moulage-based simulation training, to a control group that will receive a standard educational video on the topic of gender-based violence. This comparison will assess whether the simulation method provides better outcomes in terms of recognizing violence and improving students' attitudes.

Participants will:

Engage in a clinical simulation involving standardized patients showing signs of physical violence.

Complete pre- and post-training assessments, including attitude surveys and knowledge tests.

Reflect on their learning experience through post-intervention evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Students studying in the nursing department at Kocaeli Health and Technology University in the 2024-2025 academic year
* Registered in the Mental Health and Psychiatric Nursing course
* Accepted to participate in the study

Exclusion Criteria:

* Students not registered in the Mental Health and Psychiatric Nursing course.
* Refused to participate in the study
* Students who withdrew from the study after giving their consent.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
recognition of Physical Violence | one day
  The "Scale for Nurses and Midwives to Identify Signs of Violence Against Women" was used to define physical violence. The scale was developed to determine the knowledge levels of nurses and midwives in recognizing signs of violence against women. It consists of two sub-dimensions: "Physical Symptoms" and "Emotional Symptoms". The highest score that can be obtained from the scale is "31", the lowest score is "0". The higher the score obtained from the scale, the higher the level of knowledge about physical violence.

SECONDARY OUTCOMES:
Communication Skills | one day
  It was created by researchers by scanning the relevant literature in order to evaluate the student's communication skills with a woman who was subjected to violence during the simulation application by two observers. In the effective communication elements section; the student's face being turned towards the individual, having a relaxed posture, not having tied hands and arms, providing a private area during communication with the patient, maintaining eye contact, appearing sincere and interested, and using a soothing tone of voice are evaluated. 0-6 points can be obtained from this section. An increase in the student's score in this section indicates that he/she uses effective communication elements. In the therapeutic communication techniques section; the therapeutic communication techniques used by the student during communication are evaluated. The student is given one point for each technique he/she uses.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Health and Technology University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set: lecturer — https://kocaelisaglik.edu.tr/